CLINICAL TRIAL: NCT03840499
Title: The Role of Willingness of Participation in Cardiology Trials on the Survival of Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: Study survival - v. 1.0
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Myocardial Infarction; Chronic Heart Failure
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Willing to participate in clinical study
  Interventions: Drug: Optimal medical therapy
- Not-willing to participate in clinical study
  Interventions: Drug: Optimal medical therapy

INTERVENTIONS:
Drug: Optimal medical therapy — Optimal medical therapy

SUMMARY:
It has been shown retrospectively that participation and even the willingness improves the survival of patients after myocardial infarction or heart failure. We aimed to prospectively analyse the role of participation in cardiology trials on the survival of patients in a high volumen tertiary center.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation due to acute myocardial infarction, and or heart failure
* Singed informed consent

Exclusion Criteria:

* Previous participation in any clinical study
* Haemodinamically instable, shock, intubation
* Pregnancy, breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects hospitalised due to myocardial infarction and or heart failure.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2-years

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Heart and Vascular Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No